CLINICAL TRIAL: NCT03946059
Title: Estimating the Sensitivity of a Mobile Neuro-cognitive Platform ("BrainE") to Detect Neural Plasticity and Cognitive Enhancements Following Theta-burst Stimulation to Superior Frontal/dACC TMS Stimulation.
Brief Title: Measuring Plasticity in SFC/dACC Following Theta-Burst-Stimulation Using TMS
Acronym: BTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jyoti Mishra, Asst Professor IR, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: BrainE_TMS
Record Dates: First submitted 2019-05-07; First posted 2019-05-10 (Actual); Results first posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-02

CONDITIONS: Cognitive Control

STUDY DESIGN:
Intervention Model Description: The investigators will test the effects of two different interventions (iTBS, cTBS) on cognitive control. Each participant will receive both interventions, labeled A & B, separated a week apart.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigators will assess for each subject whether they have any guess, a priori, as to hypothesized effects of the iTBS vs. cTBS protocols (improve, impair or no change on cognition). Participant/care provider will know which stimulation is being applied (iTBS, cTBS based on labels A & B), but will not know the hypothesized effects of these two protocols. iTBS and cTBS protocols will be masked as "treatment A" and "treatment B", prior to handing the data over to PI/outcomes assessor. Analyses will thus be performed to assess whether treatment "A" or treatment "B" has an effect on cognition; and whether there are differences between these treatment protocols.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- iTBS then cTBS (Experimental): Participants in this arm first receive the iTBS brain stimulation in week 1, then have a one-week washout period and then receive cTBS brain stimulation in week 2.
  intermittent Theta-Burst-Stimulation (iTBS) entails a 2 second train of stimuli (stimuli occurring as a 50 Hz burst of three pulses separated by 200ms). Each 2 second train is followed by an 8 second pause, followed by another 2 second train. In total, 20 trains will be delivered, for a total of 200 bursts and 600 total pulses.
  continuous Theta-Burst-Stimulation (cTBS) consists of a continuous stimulus train (stimuli occurring as a 50 Hz burst of three pulses separated by 200ms). In total, 200 bursts and 600 total pulses will be delivered.
  Interventions: Device: iTBS then cTBS
- cTBS then iTBS (Experimental): Participants in this arm first receive the cTBS brain stimulation in week 1, then have a one-week washout period and then receive iTBS brain stimulation in week 2.
  Interventions: Device: cTBS then iTBS

INTERVENTIONS:
Device: iTBS then cTBS — repetitive transcranial magnetic stimulation applied with intermittent theta-burst stimulation protocol applied in week 1 and continuous theta-burst stimulation protocol applied in week 2.
  Arms: iTBS then cTBS
Device: cTBS then iTBS — repetitive transcranial magnetic stimulation applied with continuous theta-burst stimulation protocol applied in week 1 and intermittent theta-burst stimulation protocol applied in week 2.
  Arms: cTBS then iTBS

SUMMARY:
This is a study to determine whether particular forms of brain-stimulation, applied to superior frontal cortex/preSMA can affect cognition and associated frontal theta oscillations. To perform this study, the investigators first measure brain activity and cognitive performance using "BrainE", a cognitive task platform that assesses cognition on sustained attention, response inhibition, working memory, interference processing and emotion processing assessments. Next, the investigators apply brain-stimulation over a mid-frontal region associated with these tasks (mid-line frontal activity overlying superior frontal cortex/pre-SMA area). Finally, human subjects perform the "BrainE" task assessments again immediately after the brain-stimulation. The investigators compare the effects of brain stimulation on average frontal activity evoked across the cognitive tasks, and on the cognitive performance averaged across tasks. The investigators primarily compare the effects of two types of brain-stimulation against each other: intermittent Theta-Burst Stimulation (a protocol designed to excite brain activity) and continuous Theta-Burst-Stimulation (a stimulation protocol designed to inhibit brain activity).

DETAILED DESCRIPTION:
1. Brain/Behavior Recordings: to measure brain activity as described above, the investigators first ask subjects to engage in a cognitive assessment set while measuring EEG activity. For this study, the assessment set consists of the following tasks: (1) sustained attention; (2) response inhibition; (2) visuo-spatial working-memory; (3) Flanker interference processing, and (4) emotional interference processing. This battery takes about 30 minutes to complete. 24 channel EEG recordings are performed simultaneous to the cognitive tasks. Subjects perform the "BrainE" cognitive assessment, then receive brain-stimulation, and will then immediately be tested on the BrainE assessment again.
2. Brain-Stimulation: Each subject will be asked to come in twice for this study, separated by 1 week. On week one they will receive one stimulation protocol, and on the subsequent week they will receive the other (order determined randomly for each subject). The intermittent Theta-Burst-Stimulation protocol (iTBS) consists of a similar burst pattern (3 stimulation pulses 20ms apart; each burst applied every 200ms). However, after 10 bursts (2 seconds of stimulation) there is a pause for 8 seconds. 200 bursts are still applied, however due to the inter-burst intervals, this paradigm takes 200 seconds. The continuous Theta-Burst-Stimulation protocol (cTBS) consists of a burst of three stimulation pulses, applied 20ms apart; with each burst occurring every 200ms. Thus, every second participants receive 5 bursts. This continues for 40 seconds, such that participants in total receive 200 bursts or 600 pulses.

ELIGIBILITY:
Inclusion Criteria:

Adequate decisional capacity to make a choice about participating in this research study.

Exclusion Criteria:

* No major active neurologic/psychiatric disease
* No contraindications for rTMS
* No behavioral/medical factors that increase risk of seizure

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti Mishra, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- Altman Clinical & Translational Research Institute, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened for this study prior to enrollment. Any individuals with a history of seizure disorder; vascular or other lesion of the brain; administration of drugs that lower the seizure threshold; implanted or non-removable metallic objects above the neck; implanted devices with electrical circuits were excluded from enrollment.
Pre-assignment Details: No enrolled participants were excluded.
Groups:
- cTBS Then iTBS: Participants received cTBS at week 1 (1 day), washout (1 week) then iTBS at week 2 (1 day). The global cognitive task-average superior frontal theta signal was calculated as (Post - Pre)cTBS versus (Post-Pre)iTBS
- iTBS Then cTBS: Participants received iTBS at week 1 (1 day), washout (1 week) then cTBS at week 2 (1 day). The global cognitive task-average superior frontal theta signal was calculated as (Post - Pre)iTBS versus (Post-Pre)cTBS
Period: Overall Study
Arm/Group | cTBS Then iTBS | iTBS Then cTBS
Started | 13 | 12
Completed | 13 | 11
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- cTBS Then iTBS: Participants received cTBS at week 1 (1 day), washout (1 week) then iTBS at week 2 (1 day).
- iTBS Then cTBS: Participants received iTBS at week 1 (1 day), washout (1 week) then cTBS at week 2 (1 day).
- Total: Total of all reporting groups
Arm/Group | cTBS Then iTBS | iTBS Then cTBS | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 25
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 4 | 7 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 0 | 2
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Post vs. Pre Change in Mid-frontal Theta Oscillations for iTBS vs. cTBS Stimulation
Description: Change in superior frontal stimulus-evoked theta oscillations were measure on a set of cognitive tasks, specifically selective attention, response inhibition, working memory, interference processing and emotion processing tasks. The evoked EEG response (mid-frontal theta FCz as a source for superior frontal theta) was averaged across all cognitive tasks to yield a global cognitive task-averaged signal that was measured immediately before (Pre) and immediately after (Post) iTBS, and similarly immediately before (Pre) and immediately after (Post) cTBS.
Time Frame: (Post-Pre) iTBS and (Post-Pre) cTBS signals were measured one week apart.
Population: Although 25 participants enrolled, only 24 completed the study.
Measure: Mean (Standard Deviation); unit: microVolts (uV) at FCz EEG electrode
Groups:
- cTBS: Participants received cTBS intervention in one of the two study visits. The global cognitive task-average FCz theta signal was calculated as (Post-Pre)cTBS.
- iTBS: The participants received iTBS intervention in one of the two study visits. The global cognitive task-average FCz theta signal was calculated as (Post-Pre)iTBS.
Arm/Group | cTBS | iTBS
Number analyzed (Participants) | 24 | 24
microVolts (uV) at FCz EEG electrode | -0.043 (0.17) | 0.017 (0.12)

2. Secondary Outcome: Post vs. Pre Change in Cognitive Performance
Description: Change in cognitive performance was measured on a set of cognitive tasks, specifically selective attention, response inhibition, working memory, interference processing and emotion processing tasks. The cognitive performance was averaged across all cognitive tasks to yield global cognitive task-averaged performance that was measured immediately before (Pre) and immediately after (Post) iTBS, and similarly immediately before (Pre) and immediately after (Post) cTBS.
Time Frame: (Post-Pre) iTBS and (Post-Pre) cTBS cognitive performance levels were measured one week apart.
Population: Although 25 participants enrolled, only 24 completed the study.
Measure: Mean (Standard Deviation); unit: log(1/sec)
Groups:
- cTBS: Participants received cTBS intervention in one of the two study visits. The global cognitive performance was averaged across all cognitive tasks to yield global cognitive task-averaged performance that was measured immediately before (Pre) and immediately after (Post) cTBS, presented here as Post-Pre in log per second.
- iTBS: Participants received iTBS intervention in one of the two study visits. The global cognitive performance was averaged across all cognitive tasks to yield global cognitive task-averaged performance that was measured immediately before (Pre) and immediately after (Post) iTBS, presented here as Post-Pre in log per second.
Arm/Group | cTBS | iTBS
Number analyzed (Participants) | 24 | 24
log(1/sec) | 0.025 (0.027) | 0.013 (0.020)

ADVERSE EVENTS:
Time Frame: one week
Groups:
- cTBS: Participants received cTBS intervention in one of the two study visits.
- iTBS: Participants received iTBS intervention in one of the two study visits.
Arm/Group | cTBS | iTBS
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/59/NCT03946059/Prot_SAP_002.pdf